CLINICAL TRIAL: NCT02371460
Title: Maternal Omega-3 Supplementation to Reduce BronchopulmonarY Dysplasia in Very Preterm Infants (MOBYDIck Trial)
Brief Title: Maternal Omega-3 Supplementation to Reduce Bronchopulmonary Dysplasia
Acronym: MOBYDIck
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-2144, B14-09-2144-21; MOP-136964 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Bronchopulmonary Dysplasia; Child Development; Neonatal and Perinatal Conditions
Keywords: Neonatal Prematurity; Omega-3 Fatty Acids; Breastfeeding
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA-rich algal oil (Experimental): 1200mg DHA per day
  Interventions: Dietary Supplement: DHA-rich algal oil
- Placebo (Placebo Comparator): No supplementation in DHA
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: DHA-rich algal oil — Mothers will receive a DHA-rich algal oil treatment (400 mg DHA per capsule) three times a day before meals from randomization (<72 hours post-delivery) until the infant reaches 36 weeks PMA.
  Other Names: DHA group
  Arms: DHA-rich algal oil
Combination Product: Placebo — Mothers will receive a placebo capsule three times a day before meals from randomization (<72 hours post-delivery) until the infant reaches 36 weeks PMA.
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
The aim of this randomized controlled trial is to determine whether docosahexaenoic acid (or DHA, an omega-3 lipid) supplementation in lactating mothers providing breast-milk to their infant born below 29 0/7 weeks of gestational age (GA) improves BPD-free survival at 36 weeks post-menstrual age (PMA). Half of participants will receive docosahexaenoic acid (DHA), an omega-3 lipid, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Every year in Canada, 1500 babies who are born early (prematurely) develop a serious lung disease called bronchopulmonary dysplasia (BPD). BPD causes major health problems in these infants, especially in their early childhood. In most situations, breast-milk is the ideal source of nutrition for growth and development of premature babies. However, diets of Canadian mothers are generally deficient in omega-3 lipids (essential fats), resulting in lower protection from these omega-3 lipids in mother's milk-fed infants. Previous research has shown that giving DHA to mothers of premature babies is safe both for the mother and for their baby, and is an efficient way of helping babies meet their dietary requirements from breast-milk. Furthermore, this previous research also suggests that this intervention may reduce the risk of BPD in premature babies receiving breast-milk.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than or equal to 16 years
2. Pre-term delivery (230/7- 286/7 weeks gestation)
3. No contraindication to breastfeeding
4. Subject intends to provide own breast milk to infant
5. Randomization before or at 72 hours post delivery

Exclusion Criteria:

MOTHERS

1. Mother is taking > 250 mg of daily DHA supplementation for last 3 months
2. Mother who is currently enrolled or has participated in another clinical trial in which she had received an investigational drug or intervention within 3 months of the date of randomization (unless approved by the Trial Coordinating Centre)
3. Inability to comprehend and comply with study requirements
4. Participation in this study in a previous pregnancy

INFANTS

1. Significant congenital malformations in the infant (or one of the infants in case of multiple pregnancy)
2. Infant (or one of the infants in case of multiple pregnancy) who is currently enrolled in another clinical trial (unless approved by the Trial Coordinating Centre)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-06-23 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
BPD-free survival | at 36 weeks PMA
  Defined as (1- combined rate of mortality and BPD in survivors). Mortality is defined as death from any cause between randomization and 36 weeks PMA. Physiological BPD is defined as the need for oxygen and/or ventilation at 36 weeks

SECONDARY OUTCOMES:
Mortality | until 36 weeks PMA
  Mortality is defined as death from any cause.
Bronchopulmonary Dysplasia (BPD) | at 36 weeks PMA
  Physiological BPD is defined as the need for oxygen and/or ventilation at 36 weeks
Mild, moderate and severe BPD | at 36 weeks PMA
  Defined according to the severity-based National Institute of Child Health & Development (NICHD) criteria
Necrotizing enterocolitis stage 2 or greater | until first discharge home or 40 weeks PMA
  According to Bell criteria
Any intraventricular hemorrhage and severe grade III or IV | from randomization until discharge home or 40 weeks PMA
  According to Papile's classification; Screening is performed as routine care;
Periventricular leucomalacia | until discharge home or 40 weeks PMA
  Screening is performed as routine care
Sepsis | until discharge home or 40 weeks PMA
  Defined as culture-positive (blood or cerebrospinal fluid) and/or clinical infection (with antibiotics ≥5 days)
Retinopathy of prematurity (any or threshold) | until first discharge home or 40 weeks PMA
  According to the assessment by ophthalmologist, collected in the medical chart
Patent ductus arterious | until first discharge home or 40 weeks PMA
  Requiring surgical ligation
Significant cholestasis | until first discharge home or 36 weeks PMA
  Defined as conjugated serum bilirubin ≥34 µmol/L
Child anthropometry | until first discharge home or 36 weeks PMA
  Weight, length and cranial circumference as routinely measured and collected in the chart
Neuro-development | at 18-22 months corrected age (CA)
  Defined as mean cognitive, language and motor composite scores of the Bayley Scale of Infant and Toddler Development's third edition (Bayley-III)

OTHER OUTCOMES:
Supplemental Oxygen | at 36 weeks PMA
  Defined as need for supplemental oxygen (mL/min flow or FiO2)
Duration of supplemental oxygen or respiratory support | until first discharge home or 36 weeks PMA
  Defined as cumulative days on supplemental oxygen or respiratory support
Hospitalization duration | until first discharge home or 40 weeks PMA
  Defined as number of days in hospital
Cerebral palsy | at 18-22 months CA
  will be ascertained using standard definitions and severity classified using the Gross Motor Function Classification System
Child anthropometry | at 18-22 months CA
  Weight, length and cranial circumference
Deafness | until 18-22 months CA
  Hearing tests will be performed by audiologists according to standard practice
Blindness (yes/no), visual acuity +/- strabismus | until 18-22 months CA
  According to ophthalmologist or orthoptist examination
Death since 40weeks | from first discharge or 40 weeks PMA until 18-22 months CA
  Any cause
Number of hospital readmissions | From first discharge until 18-22 months CA
  Assessment by standardized interview
Respiratory morbidities | until 18-22 months CA
  Physical examination will be performed by a pediatrician and a standardized general health questionnaire (including respiratory health outcomes) will be completed. Respiratory health outcomes will include respiratory symptoms, hospital admissions for respiratory deteriorations, use of inhaled therapies.
Maternal Satisfaction | at 36 weeks PMA
  Assessment by a questionnaire
Maternal significant episodes of bleeding requiring treatment or hospitalization until 4 weeks post intervention | from date of randomization up to 40 weeks PMA
  Assessment by standardized interview
Acceptability of a study at 8 years of age involving brain magnetic resonance imaging (MRI) | at 60 months CA
  Semistructured interviews framed using the theoretical domains framework will be conducted to identify potential barriers and facilitators that may influence participation in a follow-up study with brain MRI at 8 years of age.
  A subsample of n=194 children will be eligible to participate if they have not died or withdrawn from the trial and if they were born and enrolled at the following centres:
  1. CHU de Québec-Université Laval
  2. Centre Hospitalier Universitaire de Sherbrooke, CHUS
  3. CHU Sainte-Justine
  4. Jewish General Centre
  5. McGill University Health Center, Glen Site, Montreal Children's Hospital
Child health-related quality of life | at 60 months CA
  Assessed by the Pediatric Quality of Life Inventory (PedsQL).
  A subsample of n=194 children will be eligible to participate if they have not died or withdrawn from the trial and if they were born and enrolled at the following centres:
  1. CHU de Québec-Université Laval
  2. Centre Hospitalier Universitaire de Sherbrooke, CHUS
  3. CHU Sainte-Justine
  4. Jewish General Centre
  5. McGill University Health Center, Glen Site, Montreal Children's Hospital
Behavioral problems | at 60 months CA
  Assessed by the Total Difficulties scores, Externalizing and Internalizing scores of the Strengths and Difficulties Questionnaire.
  A subsample of n=194 children will be eligible to participate if they have not died or withdrawn from the trial and if they were born and enrolled at the following centres:
  1. CHU de Québec-Université Laval
  2. Centre Hospitalier Universitaire de Sherbrooke, CHUS
  3. CHU Sainte-Justine
  4. Jewish General Centre
  5. McGill University Health Center, Glen Site, Montreal Children's Hospital
Executive function | at 60 months CA
  Assessed by the Global executive composite score of the Behavior Rating Inventory of Executive Function - Preschool.
  A subsample of n=194 children will be eligible to participate if they have not died or withdrawn from the trial and if they were born and enrolled at the following centres:
  1. CHU de Québec-Université Laval
  2. Centre Hospitalier Universitaire de Sherbrooke, CHUS
  3. CHU Sainte-Justine
  4. Jewish General Centre
  5. McGill University Health Center, Glen Site, Montreal Children's Hospital
Global developmental delay | at 60 months CA
  Assessed by the 5 developmental areas of the Ages and Stages Questionnaire.
  A subsample of n=194 children will be eligible to participate if they have not died or withdrawn from the trial and if they were born and enrolled at the following centres:
  1. CHU de Québec-Université Laval
  2. Centre Hospitalier Universitaire de Sherbrooke, CHUS
  3. CHU Sainte-Justine
  4. Jewish General Centre
  5. McGill University Health Center, Glen Site, Montreal Children's Hospital
Exposure and impact of the COVID-19 pandemic | at 60 months CA
  Impact on the home environment, quality of life, development and behavioral and executive functioning.
  A subsample of n=194 children will be eligible to participate if they have not died or withdrawn from the trial and if they were born and enrolled at the following centres:
  1. CHU de Québec-Université Laval
  2. Centre Hospitalier Universitaire de Sherbrooke, CHUS
  3. CHU Sainte-Justine
  4. Jewish General Centre
  5. McGill University Health Center, Glen Site, Montreal Children's Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Marc, MD, PhD, Principal Investigator — CHU de Québec, Université Laval; Pascal Lavoie, MD, PhD, Principal Investigator — Children's and Women's Health Centre of BC, University of British Columbia; Benoît Mâsse, PhD, Principal Investigator — CHU Sainte-Justine, Université de Montreal; Thierry Lacaze, MD, PhD, Principal Investigator — Children's Hospital of Eastern Ontario, University of Ottawa; Anne-Monique Nuyt, MD, PhD, Principal Investigator — CHU Sainte-Justine, Université de Montreal; William Fraser, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (16):
- Canada (16):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexander Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - St Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Science Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Jewish General Centre, Montreal, Quebec
  - McGill University Health Center, Glen Site, Montreal Children's Hospital, Montreal, Quebec
  - CHU de Québec-Université Laval, Centre Mère Enfant Soleil du CHUL, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marc I, Julien P, Lavoie PM. Maternal Docosahexaenoic Acid Supplementation and Bronchopulmonary Dysplasia in Infants-Reply. JAMA. 2020 Nov 24;324(20):2105. doi: 10.1001/jama.2020.19410. No abstract available. PMID 33231656
- [Background] Fougere H, Bilodeau JF, Lavoie PM, Mohamed I, Rudkowska I, Pronovost E, Simonyan D, Berthiaume L, Guillot M, Piedboeuf B, Julien P, Marc I. Docosahexaenoic acid-rich algae oil supplementation on breast milk fatty acid profile of mothers who delivered prematurely: a randomized clinical trial. Sci Rep. 2021 Nov 2;11(1):21492. doi: 10.1038/s41598-021-01017-8. PMID 34728723
- [Background] Angoa G, Pronovost E, Ndiaye ABKT, Lavoie PM, Lemyre B, Mohamed I, Simonyan D, Qureshi M, Afifi J, Yusuf K, Series T, Guillot M, Piedboeuf B, Fraser WD, Nuyt AM, Masse B, Lacaze-Masmonteil T, Marc I. Effect of Maternal Docosahexaenoic Acid Supplementation on Very Preterm Infant Growth: Secondary Outcome of a Randomized Clinical Trial. Neonatology. 2022;119(3):377-385. doi: 10.1159/000524147. Epub 2022 Apr 12. PMID 35413719
- [Background] Ndiaye ABKT, Mohamed I, Pronovost E, Angoa G, Piedboeuf B, Lemyre B, Afifi J, Qureshi M, Series T, Guillot M, Simonyan D, Yusuf K, Lavoie PM, Fraser WD, Masse B, Nuyt AM, Lacaze-Masmonteil T, Marc I. Use of SMOF lipid emulsion in very preterm infants does not affect the incidence of bronchopulmonary dysplasia-free survival. JPEN J Parenter Enteral Nutr. 2022 Nov;46(8):1892-1902. doi: 10.1002/jpen.2380. Epub 2022 May 8. PMID 35403244
- [Background] Fougere H, Greffard K, Guillot M, Rudkowska I, Pronovost E, Simonyan D, Marc I, Bilodeau JF. Docosahexaenoic acid-rich algae oil supplementation in mothers of preterm infants is associated with a modification in breast milk oxylipins profile. Lipids Health Dis. 2023 Jul 14;22(1):103. doi: 10.1186/s12944-023-01870-8. PMID 37452341
- [Background] Series T, Guillot M, Angoa G, Pronovost E, Ndiaye ABKT, Mohamed I, Simonyan D, Lavoie PM, Synnes A, Marc I; MOBYDIck trial group. Does Growth Velocity Affect Associations between Birth Weight and Neurodevelopment for Infants Born Very Preterm? J Pediatr. 2023 Sep;260:113531. doi: 10.1016/j.jpeds.2023.113531. Epub 2023 Jun 1. PMID 37268036
- [Background] Paquet SP, Pronovost E, Simonyan D, Caouette G, Matte-Gagne C, Olivier F, Bartholomew J, Morin A, Mohamed I, Marc I, Guillot M. Maternal high-dose docosahexaenoic acid supplementation and neurodevelopment at 5 Years of preterm children. Clin Nutr ESPEN. 2024 Dec;64:253-262. doi: 10.1016/j.clnesp.2024.09.029. Epub 2024 Oct 11. PMID 39396702
- [Derived] Guillot M, Synnes A, Pronovost E, Qureshi M, Daboval T, Caouette G, Olivier F, Bartholomew J, Mohamed I, Masse E, Afifi J, Hendson L, Lemyre B, Luu TM, Strueby L, Cieslak Z, Yusuf K, Pelligra G, Ducruet T, Ndiaye ABKT, Angoa G, Series T, Piedboeuf B, Nuyt AM, Fraser W, Masse B, Lacaze-Masmonteil T, Lavoie PM, Marc I. Maternal High-Dose DHA Supplementation and Neurodevelopment at 18-22 Months of Preterm Children. Pediatrics. 2022 Jul 1;150(1):e2021055819. doi: 10.1542/peds.2021-055819. PMID 35652296
- [Derived] Guillot M, Robitaille CA, Turner L, Pronovost E, Caouette G, Matte-Gagne C, Olivier F, Bartholomew J, Masse E, Morin A, Mohamed I, Marc I. Effects of maternal docosahexaenoic acid supplementation on brain development and neurodevelopmental outcomes of breastfed preterm neonates: protocol for a follow-up at preschool age of a randomised clinical trial (MOBYDIckPS). BMJ Open. 2022 May 4;12(5):e057482. doi: 10.1136/bmjopen-2021-057482. PMID 35508343
- [Derived] Marc I, Piedboeuf B, Lacaze-Masmonteil T, Fraser W, Masse B, Mohamed I, Qureshi M, Afifi J, Lemyre B, Caouette G, Bartholomew J, Nuyt AM, Julien P, Synnes A, Lucas M, Perreault T, Strueby L, Cieslak Z, Yusuf K, Pelligra G, Masse E, Larsen B, de Cabo C, Ruth C, Khurshid F, Lavoie PM. Effect of Maternal Docosahexaenoic Acid Supplementation on Bronchopulmonary Dysplasia-Free Survival in Breastfed Preterm Infants: A Randomized Clinical Trial. JAMA. 2020 Jul 14;324(2):157-167. doi: 10.1001/jama.2020.8896. PMID 32662862